CLINICAL TRIAL: NCT00833950
Title: Phase Out Treatment for Tinnitus
Brief Title: Phase Out in Tinnitus Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Prof Dr P H Van de Heyning, Antwerp University Hospital
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8/2/12
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2009-03-03 (Estimated); Status verified 2008-12

CONDITIONS: Tinnitus
Keywords: Tinnitus; Phase Out
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- narrow band noise (Experimental): Phase out in narrow band noise tinnitus patients
  Interventions: Device: Phase Out treatment in pure tone tinnitus patients

INTERVENTIONS:
Device: Phase Out treatment in pure tone tinnitus patients — Phase Out treatment: 30 min 3x/w during 6 weeks

SUMMARY:
Phase shift treatment is a new tinnitus therapy that aims at sound cancelling via complete or partial residual inhibition. This technique is based on the theory by Choy advocating that the induction of a sound wave with a 180 degree phase shift compared to the sound experienced by the patient could result in sound cancelling, likely by negation of the cortical perception of tinnitus.

The aim is to determine the efficacy of the Phase Out treatment in pure tone and narrow band noise tinnitus patients.

ELIGIBILITY:
Inclusion Criteria:

* consult ENT department UZA with tinnitus
* pure tone tinnitus or narrow band noise tinnitus
* unilateral tinnitus, or bilateral tinnitus if both ears pure tone or both ears narrow band noise
* frequency tinnitus > 1kHz
* cochlear origin tinnitus
* tinnitus duration 3 months or longer
* age 18y or more
* patient being able to cooperate
* patiënt able to fill in VAS
* normal MRI pontine angle

Exclusion Criteria:

* depression: BDI > 21
* pulsatile tinnitus
* pregnancy
* epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 3x/week

SECONDARY OUTCOMES:
Score on Tinnitus Questionnaire | week 0, week 3, week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp university Hospital, Edegem, Antwerp, Belgium